CLINICAL TRIAL: NCT01571518
Title: Optimal Timing and Duration of Daily G-CSF With Adjuvant TAC Chemotherapy in Node-positive Breast Cancer;Multicenter, Randomized, Open Label, Clinically IV Phase
Brief Title: Prevention of Neutropenia After Using G-CSF With TAC Chemotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hyuk moon Kim (Other)
Collaborators: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Hyuk moon Kim, Assistant professor, Sunchonhang University
Organization: Sunchonhang University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011-91
Record Dates: First submitted 2012-03-29; First posted 2012-04-05 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Neutropenia
Keywords: G-CSF; neutropenia; TAC
MeSH Terms: conditions — Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- early injection (Experimental): injection of G-CSF (leukostim)5㎍/kg from day 2 of TAC chemotherapy
  Interventions: Drug: late leukostim
- late injection (Sham Comparator): injection of G-CSF (leukostim)5㎍/kg from day 5 of TAC chemotherapy
  Interventions: Drug: early leukostim

INTERVENTIONS:
Drug: late leukostim — injection of G-CSF (leukostim)5㎍/kg from day 5 of TAC chemotherapy
  Other Names: 5leuko
  Arms: early injection
Drug: early leukostim — injection of G-CSF (leukostim)5㎍/kg from day 2 of TAC chemotherapy
  Other Names: 2leuko
  Arms: late injection

SUMMARY:
After resection of lymph node positive breast cancer, the injection duration and timing of Granulocyte-colony stimulating factor (G-CSF) could affect the neutropenia with TAC (Taxotere, Adriamycin, cyclophosphamide) chemotherapy.

DETAILED DESCRIPTION:
The duration and the injection timing of G-CSF are effective in the prevention of neutropenia, incidence of infection and non hematologic toxicity. With the TAC chemotherapy after resection of breast cancer, the G-CSF early injection versus late injection could change the frequency of neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* primary invasive breast carcinoma with lymph node positive with curative surgery with TAC chemotherapy

Exclusion Criteria:

* pregnancy,
* cardiovascualr disease,
* abnormal renal function,
* hematologic disorder

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
frequency of neutropenia | Change from Baseline in neutrophil count at 21days
  during the 1 cycle (21days) of ajuvant chemotherapy with TAC, record the frequency of neutropenia aftr using G-CSF (Leucostim)

CONTACTS AND LOCATIONS:
Overall Officials: Chul Wan Lim, MD,PhD, Study Chair — Soonchunhyang U Puchun Hospital
Locations (1):
- Soonchunhyang university Puchun Hospital, Puchun, South Korea

REFERENCES:
- [Result] Chan A, Fu WH, Shih V, Coyuco JC, Tan SH, Ng R. Impact of colony-stimulating factors to reduce febrile neutropenic events in breast cancer patients receiving docetaxel plus cyclophosphamide chemotherapy. Support Care Cancer. 2011 Apr;19(4):497-504. doi: 10.1007/s00520-010-0843-8. Epub 2010 Mar 17. PMID 20232087